CLINICAL TRIAL: NCT06914856
Title: Recovery Finance: Financial Health and Mental Health After Incarceration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000033658; 1R01MD018255-01 (NIH)
Record Dates: First submitted 2024-07-11; First posted 2025-04-06 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Financial Hardship; Mental Health Issue; Substance Use
Keywords: Financial Health; Incarceration; Mental Health; Substance Use
MeSH Terms: conditions — Financial Stress; Substance-Related Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Financial Capability Support (No Intervention): The participants in this arm will receive one-on-one financial coaching, which entails monthly or more frequent meetings with a financial coach. The initial meetings will be held in person and subsequent meetings may be held via zoom, phone, or in person depending on the comfort and convenience of the participant. Participants will also receive access to safe and affordable financial services, which includes support with managing any existing bank accounts, or supporting a person to open a new overdraft-free account. Coaches can also help people to access other financial products such as free tax preparation (VITA), credit builder loans, online bank accounts, or other products recommended by our Justice Tech partner.
- Financial Capability Support with Peer Support (Experimental): The participants randomized into this arm will receive services offered in the Financial Capability Support arm with the additional services of one-on-one peer support provided by a trained Recovery Support Specialist. Recovery Support Specialist, also referred to as Wellness coaches, will provide weekly meetings (30-60 minutes in duration) to the participants.
  Interventions: Behavioral: Financial Capability Support with Peer Support Services

INTERVENTIONS:
Behavioral: Financial Capability Support with Peer Support Services — The participants in this arm will receive one-on-one financial coaching, which entails monthly or more frequent meetings with a financial coach. Participants will also receive access to safe and affordable financial services, which includes support with managing any existing bank accounts, or supporting a person to open a new overdraft-free account. Coaches can also help people to access other financial products such as free tax preparation (VITA), credit builder loans, online bank accounts, or other products recommended by our Justice Tech partner. The participants will also receive will receive the additional services of one-on-one peer support provided by a trained Recovery Support Specialist. Recovery Support Specialist, also referred to as Wellness coaches, will provide weekly meetings (30-60 minutes in duration) to the participants.
  Arms: Financial Capability Support with Peer Support

SUMMARY:
This proposal will address financial wellbeing, an often overlooked but important factor impacting reentry for justice-involved people with mental health challenges, who are disproportionately Black and Latine. The project will change community level determinants by integrating financial capability support (one-on-one coaching and access to financial tools and services) into existing services and training bank and credit union staff to reduce discrimination. It will also support collaborative community efforts working towards upstream policy and legal reforms to reduce the incidence of those financial challenges.

DETAILED DESCRIPTION:
This research project will use Community Based Participatory Research (CBPR) methods to achieve the following specific aim:

1. Change community level determinants that impact financial well-being and health of the target group by training existing service provider including: i) community-based financial capability providers to be able to address financial difficulties of the target group; ii) service providers along the criminal justice pathway to be able to provide basic financial guidance to target group; iii) financial institution staff to reduce discrimination related to financial consequences of justice-involvement and mental illness. The investigator will also support community collaborations working for legal/policy reform that impacts finances of target group.
2. Use mixed methods to assess impact on community determinants, measuring integration of financial capability support into existing services, ability of financial coaches to support target group, access to financial products, attitudes, knowledge and behavior of bank staff, strength of community collaborations, and progress towards changes in laws and policies.
3. The investigator will assess impact on individuals by measuring target mechanisms (financial skills, self-efficacy and behavior) hypothesized to mediate the relationship between financial capability support and primary outcomes including financial well-being and other health determinants (employment, housing, social support, mental health supports, and belonging), secondary outcomes (health and recidivism) and mediators between primary and secondary outcomes (hope, empowerment, and mastery).
4. Assess the value of integrating peer support into community-based financial capability support for the target group by randomizing participants into two groups, financial capability support only, or financial capability support plus peer support.

ELIGIBILITY:
Inclusion Criteria:

* Have been released from jail or prison 36 months ago or less
* Self-identify as having experiences with trauma, mental illness/mental distress, or substance use
* Living or using services in the greater New Haven area
* Interested in receiving financial guidance

Exclusion Criteria:

* Less than 18 years of age
* Not have been released from jail or prison 36 months ago or less
* Not self-identify as having experiences with trauma, mental illness/mental distress, or substance use
* Not living or using services in the greater New Haven area
* Not interested in receiving financial guidance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2026-04-24 (Estimated); Study Completion 2026-04-24 (Estimated)

PRIMARY OUTCOMES:
Finances After Incarceration | Baseline Assessment, 6-Month Assessment, and 12-Month Assessment
  57 questions (plus sub-questions) measuring financial health after incarceration. Outcomes include: use of safe and affordable financial products (no/yes averaged across multiple products, range 0-1), Savings (ordinal scale for amount of savings, range 1-8), Credit score (ordinal scale for range of credit scores, range 0-6). Measuring change over time.
Money And Mental Health Scale | Baseline Assessment, 6-Month Assessment, and 12-Month Assessment
  9-item survey used to measure money and mental health, including financial well-being. Total score range is 0-4, Higher scores indicate worse effect of money on mental health. Measuring mean change over time.
Housing & Employment - QOL | Baseline Assessment, 6-Month Assessment, and 12-Month Assessment
  21-items selected from the Endicott Quality of Life measuring housing and employment. Subscales include satisfaction with living situation, satisfaction with safety, and satisfaction with work. Satisfaction rating scales range from 1-7 with higher scores indicating more satisfaction. An additional outcome is number of days worked in the last 90 days. For both satisfaction and number of days worked, measuring mean change over time.
Social Needs Screening Tool (CMS-AHC HRSN) | Baseline Assessment, 6-Month Assessment, and 12-Month Assessment
  24-item screening tool assessing social determinants of health. Outcomes include financial strain (1-3), employment help needed (1-3), living situation (1-3). Higher scores indicate more social needs. Measuring change over time.
Service Utilization | Baseline Assessment, 6-Month Assessment, and 12-Month Assessment
  31-item survey used to measure utilization of health and mental health services. Outcomes are indicated by subscales measuring number of visits to medical care outpatient, medical emergency services, mental health outpatient, mental health emergency services, psychiatric rehabilitation services, self-help programs, and alcohol/drug counseling. Other subscales indicate number of nights in a facility for a medical/surgical problem, psychiatric problem, substance use problem, or staffed residential facility. Answer formats are number of visits or days. Higher scores indicate more service use. Measuring mean change over time.
Access To Health Services (from Phenx Toolkit) | Baseline Assessment, 6-Month Assessment, and 12-Month Assessment
  10 questions measuring access to healthcare services. Outcomes include wellness visit in the past year (yes/no), delaying/missing medical care because of the cost (yes/no), number of urgent care visits, having a usual place to go for medical care (no, yes, multiple). Measuring change over time.
Intersectional Discrimination Index | Baseline Assessment, 6-Month Assessment, and 12-Month Assessment
  44-items (with branching logic) assessing discrimination, rating scales vary by question. Anticipated discrimination subscale ranges from 0-4, meaned across items. Lifetime day-to-day discrimination subscale ranges from 0-9, summed across items. Past year day-to-day discrimination subscale ranges from 0-18, summed across items. Lifetime major discrimination subscale ranges from 0-26, summed across items. Past year major discrimination subscale ranges from 0-13, summed across items. Higher scores indicate more discrimination. Measuring mean change over time.

SECONDARY OUTCOMES:
Recidivism | Baseline Assessment, 6-Month Assessment, and 12-Month Assessment
  Number of days spent in jail/prison in last 6 months. The data are assessed through self-report and the public access criminal database called ctlookup.org. Measuring mean change over time.
Wellness in 8 Dimensions Inventory | Baseline Assessment, 6-Month Assessment, and 12-Month Assessment
  67-item survey measuring wellness, rating scale 1-4, summary score meaned across items. Total score range is 1-4. Higher scores indicate higher wellness. Measuring mean change over time.
SF-12v2 (Short Form Health Survey) | Baseline Assessment, 6-Month Assessment, and 12-Month Assessment
  12-item survey measuring health, question format varies. Subscale range is 0-4 for Physical Component/Limitations Summary and Mental Component/Limitations Summary. Higher scores indicate more interference with daily living due to health problems. Measuring mean change over time.
Promis 1.0 - Anxiety for DSM-5 | Baseline Assessment, 6-Month Assessment, and 12-Month Assessment
  8-item survey measuring anxiety. Rating scale is 1-5, summary score is meaned across items. Total score range from 1-5. Higher scores indicate more anxiety. Measuring mean change over time.
Patient Health Questionnaire (PHQ-9) | Baseline Assessment, 6-Month Assessment, and 12-Month Assessment
  10-item survey measuring depression, rating scale is 0-3, summary score meaned across items. Total score ranges from 0-3. Higher scores indicating more depression. Measuring mean change over time.
PCL-5, (PTSD Checklist for DSM-5) | Baseline Assessment, 6-Month Assessment, and 12-Month Assessment
  20-item survey measuring trauma. Rating scale is 0-4, summary score meaned across items. Total score range is 0-4. Higher scores indicate more traumatic symptoms. Measuring mean change over time.
Addiction Severity Index (ASI) Limited Form | Baseline Assessment, 6-Month Assessment, and 12-Month Assessment
  37-item survey measuring addiction with higher scores indicating more addiction, question format varies. Rating scale total score range from 0-4. Total scores range 0-1 for Alcohol Use Composite Score and Drug Use Composite Score. Higher scores indicate more alcohol or drug use/problems. Measuring mean change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Annie Harper, Ph.D., Principal Investigator — Yale University; Chyrell Bellamy, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University Program for Recovery and Community Health, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via the National Data Archive (NDA).
Supporting Information: Study Protocol

DOCUMENTS (1):
  • Study Protocol (2024-03-13): https://cdn.clinicaltrials.gov/large-docs/56/NCT06914856/Prot_000.pdf